CLINICAL TRIAL: NCT06523166
Title: Direct Comparison of Cardiac CT With TEE to Evaluate Watchman FLX LAA Occluder Device Characteristics: A Multicenter Study
Brief Title: Direct Comparison of Cardiac CT With TEE to Evaluate Watchman FLX LAA Occluder Device Characteristics
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Steven Filby, MD, Physician, Interventional Cardiology, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY20231491
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Device Related Thrombosis; Peri-device Leak
Keywords: Watchman FLX; Left atrial appendage (LAA); Transesophageal echocardiography (TEE); Cardiac CTA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Left Atrial Appendage Occlusion (LAAC) with Watchman FLX. (Experimental): Patients who are status post LAAC using the Watchman FLX.
  Interventions: Procedure: Transesophageal echocardiography (TEE); Procedure: Cardiac CTA

INTERVENTIONS:
Procedure: Transesophageal echocardiography (TEE) — TEE will be performed using a 3D probe. TEE images will be acquired at the standard 0, 45, 90, and 135 degree views along with a 3D acquisition encompassing the entire LAA, device, left pulmonary vein and lateral mitral annular landmarks.
Procedure: Cardiac CTA — Cardiac CTA will be performed with ECG gating using systems with ≥ 64 detector rows and with temporal resolution that is at least 175 msec (rotation speed ≤ 350 msec for single source systems). Cardiac CTA images will be acquired for the entire cardiac cycle without ECG phase specific pulsing and with contrast appropriately timed for peak left atrial/arterial phase contrast enhancement. In addition, a targeted end systolic only delayed phase image set (45 seconds after the arterial phase scan and limited to the left atrium and appendage device) will be acquired.

SUMMARY:
The current standard of care for patients who underwent left atrial appendage closure (LAAC) is to have follow-up transesophageal echocardiogram (TEE) for device surveillance. TEE is an ultrasound of the heart done by placing a probe in the esophagus under conscious sedation. It does not use contrast but can be cumbersome to patients as it involves placing a probe in the esophagus. Cardiac computerized tomography angiography (cardiac CTA) is a non-invasive imaging modality that involves the use of certain types of x-rays, contrast (dye) and special computers to generate accurate images of the heart. Participants in this study will undergo both TEE and CTA on the same day 90 days after their LAAC procedure.

Participants will be in this research study for a period of 1 year, starting from the day of their scheduled LAAC procedure. Participants will undergo a TEE at 90 days after their procedure which is the standard of care imaging study after LAAC. As part of this study, participants will also undergo a cardiac CTA at 90 days as well. Participants will have a routine follow-up visit following device placement as per standard of care as well as a brief phone "check in" at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Subjects >18 years old planned to undergo LAAC
* eGFR ≥ 30 mL/min per 1.73 m2

Exclusion Criteria:

* Subjects below the age of 18
* non-English speaking subjects
* eGFR < 30 mL/min per 1.73 m2
* Subjects with history of contrast allergy
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
LAA patency percentage associated with peri device leak (PDL) as measured by CT scan/TEE | 3 months post procedure
LAA patency percentage associated with intra device leak (IDL) as measured by CT scan/TEE. | 3 months post procedure
LAA patency percentage associated with a combination of both PDL and IDL as measured by CT scan/TEE. | 3 months post procedure
Number of detected device-related thrombus (DRT) as measured by CT scan/TEE. | 3 months

SECONDARY OUTCOMES:
Average size of device measured in millimeters (mm) | 3 months
Percent of compression as measured by CT scan/TEE | 3 months
  Percent compression is comprised by dividing the device diameter over the device size represented as one single score.
Average depth of implant measured in millimeters (mm) | 3 months
Average hypo-attenuated thickening (HAT) measured in millimeters (mm) | 3 months
Number of adverse events as measured by medical record | Up to 7 days
  Adverse events can include respiratory failure requiring intubation or an esophageal perforation from TEE probe insertion or serious contrast related event including anaphylaxis during the CTA or acute renal failure (ARF) requiring dialysis within 7 days of the CTA.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Filby, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (5):
- United States (5):
  - Cedars Sinai, Los Angeles, California
  - St. Francis Hospital and Catholic Health, Roslyn, New York
  - Sanger Heart & Vascular Institute- Atrium Health, Charlotte, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No